CLINICAL TRIAL: NCT03885895
Title: Comparative Study for the Treatment of Freckles by Intradermal Tranexamic Acid Versus Q Switched KTP Laser (532nm)
Brief Title: Treatment of Freckles by Intradermal Tranexamic Acid Versus Q Switched KTP Laser.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Rana F Hilal, MD, Lecturer, Kasr El Aini Hospital
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: EgyFreckles
Record Dates: First submitted 2019-03-20; First posted 2019-03-22 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Therapeutic Efficacy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Participants with freckles (one side of the face) (Active Comparator): one randomized side of the face will be treated by Intradermal Tranexamic acid
  Interventions: Drug: Tranexamic Acid Injectable Product
- Participants with freckles (other side of the face) (Active Comparator): other side will be treated by Q switched KTP laser
  Interventions: Device: Q switched KTP (532nm)

INTERVENTIONS:
Drug: Tranexamic Acid Injectable Product — Ampoules used for intradermal injection
  Arms: Participants with freckles (one side of the face)
Device: Q switched KTP (532nm) — LASER
  Arms: Participants with freckles (other side of the face)

SUMMARY:
Comparative split face study in which 30 patients with freckles are recruited.One side of the face will be treated with Q Switched (QS)KTP 532nm, and the other side will be treated with intradermal tranexamic acid (TXA).

DETAILED DESCRIPTION:
One side of the face will receive QS KTPlaser at a wavelength of 532 nm, spot size 2-3 mm , power 1-1.5J/cm2 and the clinical end point is just frosting.Sessions will be every month for 2 months.

The other side of the face will be assigned to TXA intradermal microinjection in the same session using Kapron 500mg/5ml ampoules (Amoun Pharmaceutical Company), the dose of 1 ml syringe with 100mg/ml. TXA will prepared under sterile conditions. Injections will be applied intradermally on freckles area at.

The sessions of TXA will be every 2 weeks for 2 months.

Postoperatively, topical antibiotic ointment and steriod will be applied. Sunscreen then applied until the next treatment in order to minimize reactive hyperpigmentations.

Follow up after treatment monthly for 2 month.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* Age group > 18years old.

Exclusion Criteria:

* Pregnant and lactating females.
* Keloid and scarring tendancy
* Usage of invasive or semi invasive procedures for treatment of freckles such as chemical peeling , dermaroller..etc. 2 months prior to the study.
* Oral Isotretinoin 6 months prior to the study.
* Active herpetic lesions.
* Any concurrent active skin disease within the treated area.
* Photosensitive skin conditions such as systemic lupus erythematous.
* History of delayed wound healing.
* Bleeding diathesis.
* Medical conditions such as autoimmune diseases.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Pigmentation and severity index by clinical evaluation | 6 months to 1 year
  Evaluate efficacy of intradermal tranexamic acid versus Q switched KTP laser in the treatment of freckles before treatment, after treatment and after follow-up
Melanin Index change by spectrophotometer | 6 months to 1 year
  Evaluate efficacy of intradermal tranexamic acid versus Q switched KTP laser in the treatment of freckles before treatment, after treatment and after follow-up
Blinded observers' evaluation | 6 months to 1 year
  Evaluate efficacy of intradermal tranexamic acid versus Q switched KTP laser in the treatment of freckles before treatment, after treatment and after follow-up
Patient satisfaction rate | 6 months to 1 year
  Evaluate efficacy of intradermal tranexamic acid versus Q switched KTP laser in the treatment of freckles before treatment, after treatment and after follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr El Ainy university hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No